CLINICAL TRIAL: NCT00399802
Title: A Phase II Study to Assess the Safety, Tolerability, and Efficacy of MK-0822 (Cathepsin-K Inhibitor) in the Treatment of Women With Breast Cancer and Established Bone Metastases (MBD)
Brief Title: A Study to Examine the Effects of an Experimental Drug on Women With Breast Cancer and Metastatic Bone Disease (MBD)(0822-016)(COMPLETED)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0822-016; 2006_533 (Other: Merck Registration Number); MK-0822-016 (Other: Merck Protocol Number)
Record Dates: First submitted 2006-11-14; First posted 2006-11-15 (Estimated); Results first posted 2018-02-01 (Actual); Last update posted 2018-08-16 (Actual); Status verified 2018-07

CONDITIONS: Breast Cancer; Metastatic Bone Disease
MeSH Terms: conditions — Breast Neoplasms; Bone Diseases | interventions — Zoledronic Acid; odanacatib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Single IV infusion of ZA 4 mg (Active Comparator): Participants will receive a single IV infusion of ZA 4 mg at the start of treatment and a once-daily odanacatib matching placebo tablet for 4 weeks.
  Interventions: Drug: ZA; Drug: Odanacatib matching placebo
- Odanacatib 5 mg (Experimental): Participants will receive a once-daily odanacatib 5 mg tablet for 4 weeks and a single IV infusion of ZA matching placebo at the start of treatment.
  Interventions: Drug: Odanacatib; Drug: ZA matching placebo

INTERVENTIONS:
Drug: ZA — Single ZA 4 mg IV infusion at the start of treatment
  Other Names: Zometa®
  Arms: Single IV infusion of ZA 4 mg
Drug: Odanacatib — Once-daily odanacatib 5 mg tablet for 4 weeks
  Other Names: MK-0822
  Arms: Odanacatib 5 mg
Drug: Odanacatib matching placebo — Once-daily odanacatib matching placebo for 4 weeks
  Arms: Single IV infusion of ZA 4 mg
Drug: ZA matching placebo — Single IV infusion of ZA matching placebo given at the start of treatment
  Arms: Odanacatib 5 mg

SUMMARY:
This is a 4-week study to examine the effects of a new experimental medication on women with breast cancer and established bone metastases. This study will enroll approximately 45 women. The primary hypotheses are: (1) odanacatib will result in a substantial suppression of urinary N-telopeptide of type I collagen (u-NTx) similar to that achieved with an intravenous (IV) infusion of zoledronic acid (ZA) over 4 weeks of treatment; and (2) odanacatib (MK-0822) will be safe and well tolerated during 4 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patient has histologically or cytologically-confirmed breast cancer
* Patient has documented skeletal metastases

Exclusion Criteria:

* Patient is undergoing current oral bisphosphonate therapy, or has a history of oral bisphosphonate use within 6 months of entry into study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2006-11-16 (Actual); Primary Completion 2007-12-05 (Actual); Study Completion 2007-12-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Jensen AB, Wynne C, Ramirez G, He W, Song Y, Berd Y, Wang H, Mehta A, Lombardi A. The cathepsin K inhibitor odanacatib suppresses bone resorption in women with breast cancer and established bone metastases: results of a 4-week, double-blind, randomized, controlled trial. Clin Breast Cancer. 2010 Dec 1;10(6):452-8. doi: 10.3816/CBC.2010.n.059. PMID 21147688

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Intravenous (IV) Infusion of Zoledronic Acid (ZA) 4 mg: Participants received a single IV infusion of ZA 4 mg at the start of treatment and a once-daily odanacatib matching placebo tablet for 4 weeks.
- Once-daily Odanacatib 5 mg: Participants received a once-daily odanacatib 5 mg tablet for 4 weeks and a single IV infusion of ZA matching placebo at the start of treatment.
Period: Overall Study
Arm/Group | Single Intravenous (IV) Infusion of Zoledronic Acid (ZA) 4 mg | Once-daily Odanacatib 5 mg
Started | 14 | 29
Completed | 14 | 26
Not Completed | 0 | 3
Not completed — Adverse Event | 0 | 2
Not completed — Participant discontinued by mistake | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Single IV Infusion of ZA 4 mg: Participants received a single IV infusion of ZA 4 mg at the start of treatment and a once-daily odanacatib matching placebo tablet for 4 weeks.
- Total: Total of all reporting groups
Arm/Group | Single IV Infusion of ZA 4 mg | Once-daily Odanacatib 5 mg | Total
Number analyzed (Participants) | 14 | 29 | 43
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.3 (8.3) | 59.4 (10.2) | 59.7 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 29 | 43
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change From Baseline in Urinary N-telopeptide of Type I Collagen (u-NTx) at Week 4
Description: u-NTx is a biochemical index of bone resorption. Participants provided urine specimens on Day 1 (baseline) and at Week 4 for measurement of u-NTx.
Time Frame: Baseline and Week 4
Population: All randomized participants who took at least one dose of study drug and had available u-NTx data for Baseline and Week 4
Measure: Mean (95% Confidence Interval); unit: Percentage change
Arm/Group | Single IV Infusion of ZA 4 mg | Once-daily Odanacatib 5 mg
Number analyzed (Participants) | 14 | 27
Percentage change | -73 [-80 to -62] | -77 [-82 to -71]

2. Primary Outcome: Number of Participants Who Experienced an Adverse Event (AE)
Description: An AE is defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a study drug, whether or not it is considered related to the study drug.
Time Frame: Up to 6 weeks
Population: All randomized participants who took at least one dose of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Single IV Infusion of ZA 4 mg | Once-daily Odanacatib 5 mg
Number analyzed (Participants) | 14 | 29
Participants | 10 | 20

3. Primary Outcome: Number of Participants Who Discontinued Treatment Due to an AE
Description: as for outcome 2
Time Frame: Up to 4 weeks
Population: All randomized participants who took at least one dose of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Single IV Infusion of ZA 4 mg | Once-daily Odanacatib 5 mg
Number analyzed (Participants) | 14 | 29
Participants | 0 | 2

4. Secondary Outcome: Percentage Change From Baseline in Urinary Deoxypyridinoline (u-DPD) at Week 4
Description: u-DPD is a biochemical marker of bone resorption. Participants provided urine specimens on Day 1 (baseline) and Week 4 for measurement of u-DPD.
Time Frame: Baseline and Week 4
Population: All randomized participants who took at least one dose of study drug and had available u-DPD data for Baseline and Week 4
Measure: Mean (95% Confidence Interval); unit: Percentage change
Arm/Group | Single IV Infusion of ZA 4 mg | Once-daily Odanacatib 5 mg
Number analyzed (Participants) | 13 | 27
Percentage change | -52 [-64 to -36] | -30 [-43 to -15]

ADVERSE EVENTS:
Time Frame: Up to 6 weeks
Description: All randomized participants who took at least one dose of study drug
Arm/Group | Single IV Infusion of ZA 4 mg | Once-daily Odanacatib 5 mg
Serious Adverse Events (participants affected / at risk) | 2/14 | 4/29
Other Adverse Events (participants affected / at risk) | 10/14 | 17/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single IV Infusion of ZA 4 mg (N=14) | Once-daily Odanacatib 5 mg (N=29)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single IV Infusion of ZA 4 mg (N=14) | Once-daily Odanacatib 5 mg (N=29)
Palpitations (Cardiac disorders) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (5) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 5 (5)
Asthenia (General disorders) | 0 (0) | 2 (3)
Chills (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (2) | 1 (1)
Oedema (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Herpes virus infection (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 1 (1)
Blood calcium decreased (Investigations) | 1 (1) | 0 (0)
Blood sodium decreased (Investigations) | 1 (1) | 0 (0)
Haematocrit decreased (Investigations) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 4 (8) | 6 (11)
Metamyelocyte count increased (Investigations) | 1 (1) | 0 (0)
Monocyte count increased (Investigations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0)
Red blood cell count decreased (Investigations) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 1 (1) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (4)
Bone pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 2 (3)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 4 (5)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Phlebitis (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The SPONSOR must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the SPONSOR as confidential must be deleted prior to submission.